CLINICAL TRIAL: NCT03377907
Title: Perioperative Pain Alleviation of Forearm Fractures Using a Combination of Hematoma Block and Intravenous Regional Anesthesia by Ketamine and Lidocaine
Brief Title: Pain Alleviation of Forearm Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed mamdouh mohammed mahmoud, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB17100203
Record Dates: First submitted 2017-12-12; First posted 2017-12-19 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Pain; Forearm Fracture
Keywords: IVRA; hematoma block
MeSH Terms: conditions — Pain | interventions — Ketamine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ketamine in hematoma block (Active Comparator): Ketamine used in hematoma block
  Interventions: Drug: ketamine in hematoma block
- ketamine intravenous anesthesia (Active Comparator): ketamine used in local intravenous anesthesia
  Interventions: Drug: ketamine in local intravenous anesthesia
- lidocaine intravenous anesthesia (Active Comparator): 2.5 mg/kg of lidocaine 2% diluted with saline to a total volume of 40 ml.
  Interventions: Drug: Lidocaine Hydrochloride

INTERVENTIONS:
Drug: ketamine in hematoma block — ketamine used in local hematoma block only
  Arms: Ketamine in hematoma block
Drug: ketamine in local intravenous anesthesia — ketamine will be used with lidocaine in local intravenous anesthesia
  Arms: ketamine intravenous anesthesia
Drug: Lidocaine Hydrochloride — 2.5 mg/kg of lidocaine 2% in intravenous regional anesthesia
  Arms: lidocaine intravenous anesthesia

SUMMARY:
fractures of upper limb induce much pain . A lot of modalities are available to alleviate pain. fracture hematoma block, and intravenous regional anesthesia seem to be cost effective and attractive options

DETAILED DESCRIPTION:
Fractures of the forearm are extremely common, Pain relief is of utmost importance in forearm fractures which may need manipulation immediately for reduction followed by operative intervention

The characteristic features of ideal analgesia during reduction are determined by safety, simplicity, affectivity and costs. Giventhe logistic difficulty of providing such anesthesia to such large number of patients simpler alternatives to conventional anesthesia have been tried. Hematoma Block alone, Hematoma Block with sedation, Bier's Block (Intravenous regional anesthesia), regional nerve blocks, sedation have been compared to general anesthesia to evaluate the efficacy, effectiveness, safety in treating such patients

Amongst various techniques, HB and IVRA are attractive options. However, while HB has been demonstrated to be safe simple and has been used effectively for treatment of radius fractures in ER and for immediate pain relief it doesn't provide muscular relaxation and may not be sufficient for any operative intervention

IVRA is suitable for operations of the distal extremities, in situations where it is safe and easy to apply an occlusive tourniquet. The primary advantages of IVRA are its simplicity, reliability, and cost-effectiveness. . It is a regional anesthetic technique that is easy to perform, with success rates varying between 94% and 98%.For these reasons, it remains a popular choice among anesthesiologists.

A combination of blocks is usually done to overcome the deficiencies of individual blocks and to improve operating conditions or to prolong post operative analgesia. However the use of dual technique of IVRA and HB with local anesthetic only offered near absence of post operative analgesia

Lidocaine is the most frequently used LA for IVRA and HB

Different agents have been used as additive to local anesthetic for IVRA including phencyclidines, non-steroidal anti inflammatory drugs, opioids, and muscle relaxants. Ketamine is an effective anesthetic agent for IVRA at concentrations between 0.3% and 0.5%.it improves quality of anesthesia and peri operative analgesia without causing side effects

Ketamine, a phenyl-piper dine derivative, was first synthesized in the early 1960 as an IV anesthetic agent. At sub anesthetic doses, ketamine exerts a noncompetitive blockade of N -methyl aspartate (NMDA) receptors. NMDA receptors play a major role in synaptic plasticity and are specifically implicated in central nervous system facilitation of pain processing. NMDA receptor antagonists have been implicated in perioperative pain management. Ketamine also has local anesthetic qualities, which have been studied as a sole agent for IVRA. In addition to spinal cord NMDA receptors, NMDA receptors have also been identified on peripheral unmyelinated sensory axons. This can explain why ketamine as an NMDA receptor antagonist was able to attenuate the tourniquet pain.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged more than 18 years old.
* American Society of Anesthesiologists (ASA) physical status I or II.
* Patients scheduled for closed fracture of distal upper extremity within 7 days, requiring open or closed reduction and internal fixation.
* Patients scheduled for procedure lasting less than 90 minutes.

Exclusion Criteria:

* Patients having cardiovascular co-morbidities.
* Compound or contaminated fracture.
* Peripheral vascular disease, sickle cell disease or coagulation disorders.
* Allergy to the local anesthetics or to the drugs used in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
pain assessment | 24 hours
  pain will be assessed by numerical rating scale

SECONDARY OUTCOMES:
analgesia requirement | 24 hours
  time of first analgesia requirement

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Egypt